CLINICAL TRIAL: NCT00003126
Title: A Randomized Controlled Phase III Adjuvant Trial of High-Dose Bolus IL-2 in Patients With High-Risk Renal Cell Carcinoma
Brief Title: Interleukin-2 in Treating Patients With Stage III or Stage IV Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 852006
Record Dates: First submitted 1999-11-01; First posted 2003-10-28 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Cancer
Keywords: renal cell cancer; renal cell carcinoma; interleukin-2
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin-2 (IL-2) (Experimental): Patients randomized to this arm will receive one course of IL-2 [600,000 U/kg every 8 hours on post-operative days 1 to 5 and days 15 to 19 (maximum 28 doses)].
  Interventions: Drug: Interleukin-2
- Observation (No Intervention): Patients randomized to this arm will receive their normal medical care

INTERVENTIONS:
Drug: Interleukin-2 — High-dose bolus interleukin-2 is a systemic therapy used to treat metastatic RCC
  Other Names: IL-2; Aldesleukin
  Arms: Interleukin-2 (IL-2)

SUMMARY:
The purpose of this study is to assess the efficacy of post-operative high-dose bolus interleukin-2 (IL-2) in patients with high-risk renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
The primary objective of this prospective, randomized, controlled trial is to compare the disease-free and overall survival of patients with stage III or IV high-risk renal cell carcinoma (RCC) who were treated with adjuvant high-dose interleukin-2 vs observation alone.

Patients are stratified according to their disease classification and randomized to one course of IL-2 [600,000 U/kg every 8 hours on days 1 to 5 and days 15 to 19 (maximum 28 doses)] or observation.

ELIGIBILITY:
Inclusion Criteria

* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function as defined by a white blood cell (WBC) count of 4,000/L; a platelet count of 100,000/L; a Hemoglobin level of 10 g/dL; a serum creatinine of 1.5 mg/dL or creatinine clearance of 60 mL/min; and a direct bilirubin level of 1.5 mg/dL.
* Forced expiratory volume at 1 second more than 2.0 L or 75% of predicted for height and age from pre-enrollment pulmonary function testing.
* No history or evidence of cardiac disease on ECG
* No prior systemic treatment for RCC, but patients may have received prior locoregional radiation therapy to solitary resectable metastases, which must have undergone surgical resection before enrollment.
* No prior history of invasive malignancy in the past 5 years
* Human immunodeficiency virus (HIV) negative
* Female patients must not be pregnant or planning to become pregnant

Exclusion criteria

• Age younger than 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1997-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 60 months
  Disease free survival will be compared between the two cohorts (i.e., IL-2 versus Observation). Time will be calculated as the difference in months from date of treatment to date of death or recurrence (whichever occurs first). Patients remaining disease-free will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Overall survival | 60 months
  Overall survival will be compared between the two cohorts (i.e., IL-2 versus Observation). Time will be calculated as the difference in months from date of treatment to date of death. Living patients will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I. Clark, MD, Principal Investigator — Loyola University
Locations (15):
- United States (15):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Summit Medical Center, Oakland, California
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Jemal A, Murray T, Samuels A, Ghafoor A, Ward E, Thun MJ. Cancer statistics, 2003. CA Cancer J Clin. 2003 Jan-Feb;53(1):5-26. doi: 10.3322/canjclin.53.1.5. PMID 12568441
- [Background] Skinner DG, Colvin RB, Vermillion CD, Pfister RC, Leadbetter WF. Diagnosis and management of renal cell carcinoma. A clinical and pathologic study of 309 cases. Cancer. 1971 Nov;28(5):1165-77. doi: 10.1002/1097-0142(1971)28:53.0.co;2-g. No abstract available. PMID 5125665
- [Background] Robson CJ, Churchill BM, Anderson W. The Results of Radical Nephrectomy for Renal Cell Carcinoma. J Urol. 2017 Feb;197(2S):S111-S113. doi: 10.1016/j.juro.2016.10.095. Epub 2016 Dec 21. No abstract available. PMID 28012766
- [Background] Motzer RJ, Mazumdar M, Bacik J, Berg W, Amsterdam A, Ferrara J. Survival and prognostic stratification of 670 patients with advanced renal cell carcinoma. J Clin Oncol. 1999 Aug;17(8):2530-40. doi: 10.1200/JCO.1999.17.8.2530. PMID 10561319
- [Background] Messing EM, Manola J, Wilding G, Propert K, Fleischmann J, Crawford ED, Pontes JE, Hahn R, Trump D; Eastern Cooperative Oncology Group/Intergroup trial. Phase III study of interferon alfa-NL as adjuvant treatment for resectable renal cell carcinoma: an Eastern Cooperative Oncology Group/Intergroup trial. J Clin Oncol. 2003 Apr 1;21(7):1214-22. doi: 10.1200/JCO.2003.02.005. PMID 12663707
- [Background] Poster DS, Bruno S, Penta JS, Pinna K, Vilk P, Macdonald JS. Current status of chemotherapy, hormonal therapy, and immunotherapy in the treatment of renal cell carcinoma. Am J Clin Oncol. 1982 Feb;5(1):53-60. PMID 7081138
- [Background] Finney R. The value of radiotherapy in the treatment of hypernephroma--a clinical trial. Br J Urol. 1973 Jun;45(3):258-69. doi: 10.1111/j.1464-410x.1973.tb12152.x. No abstract available. PMID 4712834
- [Background] Kjaer M, Frederiksen PL, Engelholm SA. Postoperative radiotherapy in stage II and III renal adenocarcinoma. A randomized trial by the Copenhagen Renal Cancer Study Group. Int J Radiat Oncol Biol Phys. 1987 May;13(5):665-72. doi: 10.1016/0360-3016(87)90283-5. PMID 3553111
- [Background] Naito S, Kumazawa J, Omoto T, Iguchi A, Sagiyama K, Osada Y, Hiratsuka Y. Postoperative UFT adjuvant and the risk factors for recurrence in renal cell carcinoma: a long-term follow-up study. Kyushu University Urological Oncology Group. Int J Urol. 1997 Jan;4(1):8-12. doi: 10.1111/j.1442-2042.1997.tb00130.x. PMID 9179659
- [Background] Pizzocaro G, Piva L, Colavita M, Ferri S, Artusi R, Boracchi P, Parmiani G, Marubini E. Interferon adjuvant to radical nephrectomy in Robson stages II and III renal cell carcinoma: a multicentric randomized study. J Clin Oncol. 2001 Jan 15;19(2):425-31. doi: 10.1200/JCO.2001.19.2.425. PMID 11208835
- [Background] Rosenberg SA, Yang JC, Topalian SL, Schwartzentruber DJ, Weber JS, Parkinson DR, Seipp CA, Einhorn JH, White DE. Treatment of 283 consecutive patients with metastatic melanoma or renal cell cancer using high-dose bolus interleukin 2. JAMA. 1994 Mar 23-30;271(12):907-13. PMID 8120958
- [Background] Fyfe G, Fisher RI, Rosenberg SA, Sznol M, Parkinson DR, Louie AC. Results of treatment of 255 patients with metastatic renal cell carcinoma who received high-dose recombinant interleukin-2 therapy. J Clin Oncol. 1995 Mar;13(3):688-96. doi: 10.1200/JCO.1995.13.3.688. PMID 7884429
- [Background] Fisher RI, Rosenberg SA, Fyfe G. Long-term survival update for high-dose recombinant interleukin-2 in patients with renal cell carcinoma. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S55-7. PMID 10685660
- [Background] Margolin KA, Rayner AA, Hawkins MJ, Atkins MB, Dutcher JP, Fisher RI, Weiss GR, Doroshow JH, Jaffe HS, Roper M, et al. Interleukin-2 and lymphokine-activated killer cell therapy of solid tumors: analysis of toxicity and management guidelines. J Clin Oncol. 1989 Apr;7(4):486-98. doi: 10.1200/JCO.1989.7.4.486. PMID 2647914
- [Background] Belldegrun A, Webb DE, Austin HA 3rd, Steinberg SM, White DE, Linehan WM, Rosenberg SA. Effects of interleukin-2 on renal function in patients receiving immunotherapy for advanced cancer. Ann Intern Med. 1987 Jun;106(6):817-22. doi: 10.7326/0003-4819-106-6-817. PMID 3495213
- [Background] Atkins MB, Sparano J, Fisher RI, Weiss GR, Margolin KA, Fink KI, Rubinstein L, Louie A, Mier JW, Gucalp R, et al. Randomized phase II trial of high-dose interleukin-2 either alone or in combination with interferon alfa-2b in advanced renal cell carcinoma. J Clin Oncol. 1993 Apr;11(4):661-70. doi: 10.1200/JCO.1993.11.4.661. PMID 8478661
- [Background] Weiss GR, Margolin KA, Aronson FR, Sznol M, Atkins MB, Dutcher JP, Gaynor ER, Boldt DH, Doroshow JH, Bar MH, et al. A randomized phase II trial of continuous infusion interleukin-2 or bolus injection interleukin-2 plus lymphokine-activated killer cells for advanced renal cell carcinoma. J Clin Oncol. 1992 Feb;10(2):275-81. doi: 10.1200/JCO.1992.10.2.275. PMID 1732429
- [Background] Atkins MB, Dutcher J, Weiss G, Margolin K, Clark J, Sosman J, Logan T, Aronson F, Mier J; Cytokine Working Group. Kidney cancer: the Cytokine Working Group experience (1986-2001): part I. IL-2-based clinical trials. Med Oncol. 2001;18(3):197-207. doi: 10.1385/MO:18:3:197. PMID 11917944
- [Background] Guinan P, Sobin LH, Algaba F, Badellino F, Kameyama S, MacLennan G, Novick A. TNM staging of renal cell carcinoma: Workgroup No. 3. Union International Contre le Cancer (UICC) and the American Joint Committee on Cancer (AJCC). Cancer. 1997 Sep 1;80(5):992-3. doi: 10.1002/(sici)1097-0142(19970901)80:53.0.co;2-q. No abstract available. PMID 9307205
- [Background] Dutcher J, Atkins MB, Margolin K, Weiss G, Clark J, Sosman J, Logan T, Aronson F, Mier J; Cytokine Working Group. Kidney cancer: the Cytokine Working Group experience (1986-2001): part II. Management of IL-2 toxicity and studies with other cytokines. Med Oncol. 2001;18(3):209-19. doi: 10.1385/MO:18:3:209. PMID 11917945
- [Background] Upton MP, Parker RA, Youmans A, McDermott DF, Atkins MB. Histologic predictors of renal cell carcinoma response to interleukin-2-based therapy. J Immunother. 2005 Sep-Oct;28(5):488-95. doi: 10.1097/01.cji.0000170357.14962.9b. PMID 16113605
- [Background] Negrier S, Escudier B, Lasset C, Douillard JY, Savary J, Chevreau C, Ravaud A, Mercatello A, Peny J, Mousseau M, Philip T, Tursz T. Recombinant human interleukin-2, recombinant human interferon alfa-2a, or both in metastatic renal-cell carcinoma. Groupe Francais d'Immunotherapie. N Engl J Med. 1998 Apr 30;338(18):1272-8. doi: 10.1056/NEJM199804303381805. PMID 9562581
- [Background] McDermott DF, Regan MM, Clark JI, Flaherty LE, Weiss GR, Logan TF, Kirkwood JM, Gordon MS, Sosman JA, Ernstoff MS, Tretter CP, Urba WJ, Smith JW, Margolin KA, Mier JW, Gollob JA, Dutcher JP, Atkins MB. Randomized phase III trial of high-dose interleukin-2 versus subcutaneous interleukin-2 and interferon in patients with metastatic renal cell carcinoma. J Clin Oncol. 2005 Jan 1;23(1):133-41. doi: 10.1200/JCO.2005.03.206. PMID 15625368
- [Background] Dutcher JP, Logan T, Gordon M, Sosman J, Weiss G, Margolin K, Plasse T, Mier J, Lotze M, Clark J, Atkins M. Phase II trial of interleukin 2, interferon alpha, and 5-fluorouracil in metastatic renal cell cancer: a cytokine working group study. Clin Cancer Res. 2000 Sep;6(9):3442-50. PMID 10999727
- [Result] Clark JI, Atkins MB, Urba WJ, Creech S, Figlin RA, Dutcher JP, Flaherty L, Sosman JA, Logan TF, White R, Weiss GR, Redman BG, Tretter CP, McDermott D, Smith JW, Gordon MS, Margolin KA. Adjuvant high-dose bolus interleukin-2 for patients with high-risk renal cell carcinoma: a cytokine working group randomized trial. J Clin Oncol. 2003 Aug 15;21(16):3133-40. doi: 10.1200/JCO.2003.02.014. Epub 2003 Jun 16. PMID 12810695